CLINICAL TRIAL: NCT01573377
Title: Efficacy of Metformin and Diane-35 on PCOS Patients,a Randomized, Controlled, Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-Qifu Li
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: polycystic ovary syndrome; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin; Ethinyl Estradiol; Cyproterone Acetate; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental): 425mg bid for morning and evening after meals, one week after treatment, increase the dosage to 850 mg bid. If the patients have side effects such as nausea, diarrhea and other gastrointestinal symptoms, the dose would be reduced to 425mg bid for 1 week, and try the dosage to 425mg tid again, until the maximum tolerated dose.
  Interventions: Drug: Metformin
- Ethinylestradiol and Cyproterone Acetate (Experimental): From the first day of the menstruation, oral administration of one pill daily for 21 days consecutively, then discontinue using the pill for seven days, and on the eighth day, restart taking the pill.
  Interventions: Drug: Ethinylestradiol and Cyproterone Acetate

INTERVENTIONS:
Drug: Metformin — 425mg bid for morning and evening after meals, one week after treatment, increase the dosage to 850 mg bid. If the patients have side effects such as nausea, diarrhea and other gastrointestinal symptoms, the dose would be reduced to 425mg bid for 1 week, and try the dosage to 425mg tid again, until the maximum tolerated dose.
  Other Names: Glucophage
  Arms: metformin
Drug: Ethinylestradiol and Cyproterone Acetate — from the first day of bleeding of the menstrual cycle, daily oral administration of one pill for 21 days consecutively, then stopped taking the pill for seven days, and on the eighth day to start taking the pill again.
  Other Names: Diane-35
  Arms: Ethinylestradiol and Cyproterone Acetate

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrinopathies in reproductive-age women, and it affects 5-7% of this group. It is characterized by disturbed menstrual cycle, ovulatory dysfunction and hyperandrogenism. Over 40% of PCOS women might become the patients with impaired glucose tolerance or type 2 diabetes. It has been confirmed that insulin resistance (IR) is a common feature in PCOS and adipokines might play roles in the pathogenesis of IR and PCOS, because these adipokines have wide-ranging effects on carbohydrate and lipid metabolism.

The present clinical trial intends to compare the effects of metformin and oral contraceptives on PCOS patients, focusing on the insulin sensitivity, ovulation, and menstrual cycle etc. The investigators also aim to study the effects of metformin on serum adipokine levels(such as pigment epithelium-derived factor, progranulin etc.)in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

with at least two of the following features : (i) oligo-amenorrhea or chronic anovulation; (ii) clinical and/or biochemical hyperandrogenism; (iii) ultrasound appearance of polycystic ovaries

Exclusion Criteria:

- other known causes of hyperandrogenemia and ovulatory dysfunction, including 21-hydroxylase deficiency, congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumors, thyroid disease, and hyperprolactinemia.

use of hormone medications (including oral contraceptives) within the past month and the use of medicines that affect insulin sensitivity (e.g., metformin or thiazolidinediones) within the past three months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
the efficacy of Metformin and Diane-35 | at 12 weeks
  Ovulation,Menstrual cycle,Insulin sensitivity

SECONDARY OUTCOMES:
changes of adipokine（PEDF,GPRN，etc）levels from baseline | at 12 weeks
  changes of adipokine（PEDF,GPRN，etc）levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China